CLINICAL TRIAL: NCT00852930
Title: Low Level Laser Treatment and Breast Cancer Related Lymphedema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sheila Ridner, professor, Vanderbilt University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 090118
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema
Keywords: lymphedema; quality of life; breast cancer; symptoms; lymphedema in breast cancer survivors
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Lasers; Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- laser alone (Experimental): The intervention was therapist administered low level laser therapy using low level laser, number of sessions based upon patient response
  Interventions: Procedure: laser alone
- mld alone (Active Comparator): The intervention was therapist administered manual lymphatic drainage (mld) using standard massage techniques,number of sessions based upon patient response
  Interventions: Procedure: manual lymphatic drainage
- laser and mld combined (Experimental): The intervention was therapist administered low level laser and mld using low level laser and standard massage techniques, number of sessions based upon patient response
  Interventions: Procedure: laser and MLD combined

INTERVENTIONS:
Procedure: laser and MLD combined — The intervention is therapist administered laser and mld treatment combined
  Arms: laser and mld combined
Procedure: laser alone — The intervention is therapist administered laser
  Arms: laser alone
Procedure: manual lymphatic drainage — The intervention is therapist administered manual lymphatic drainage
  Arms: mld alone

SUMMARY:
Manual Lymphatic Drainage (massage therapy) with compression (wearing a tight sleeve on the arm) is the current standard of treatment for breast cancer related lymphedema (arm swelling). Low-Level Laser Therapy (LLLT) was approved in 2006 by the FDA for professional and self/home treatment of lymphedema. LLLT is being offered as a treatment option in many lymphedema treatment settings, but there are few studies of the effectiveness of LLLT as a stand-alone lymphedema treatment or as a possible complementary lymphedema treatment modality to Manual Lymphatic Drainage. The objective of this proposed pilot study is to examine the impact of Advance Practice Nurse (ANP) administered LLLT, as both a stand-alone and complementary treatment, on arm volume, symptoms, and quality of life (QOL) in breast cancer survivors with lymphedema. Findings from this pilot study will be used to determine if LLLT has possible value in the treatment of lymphedema and warrants subsequent evaluation in a larger study.

DETAILED DESCRIPTION:
The purpose of this proposed pilot study is to examine the impact of Advance Practice Nurse (ANP) administered LLLT, as both a stand-alone and complementary treatment, on arm volume, symptoms, and quality of life (QOL) in breast cancer survivors with related LE. Findings from this pilot randomized study will be used to determine if LLLT has possible value in the treatment of LE and warrants subsequent evaluation in a larger study.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer survivors will be included if they:

1. are age 21 or older;
2. require professional treatment for Stage I or II lymphedema as defined by the International Society of Lymphology;
3. have an order for lymphedema treatment; and
4. are willing and able to drive to the study sites.

Exclusion Criteria:

Individuals will not be included if they:

1. are actively undergoing intravenous chemotherapy or radiation therapy;
2. have a history of bilateral lymphedema that prohibits extracellular fluid comparison to an unaffected limb;
3. are unable to stand upright for measurement of height and weight;
4. have active/metastatic cancer;
5. are pregnant,:
6. have artificial joints in areas where electrode placement is critical, or have a pacemaker/internal defibrillator; or
7. have congestive heart failure (CHF), chronic/acute renal or hepatic disease, pulmonary edema, thrombophlebitis, deep vein thrombosis (DVT), acute infection of any kind, and inflammation in the trunk or arms.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sheila h ridner, phd, Principal Investigator — Vanderbilt Univeristy
Locations (1):
- Vanderbilt University School of Nursing, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Therapy Alone: therapist administered laser treatment
  laser: therapist administered laser
- Mld Alone: therapist administered manual lymphatic drainage
  manual lymphatic drainage: therapist administered massage therapy
- Laser and Mld Combined: therapist administered laser and mld
  Low Level Laser Therapy with Manual Lymphatic Drainage: therapist will give both mld and laser treatment
Period: Overall Study
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Started | 16 | 17 | 17
Completed | 15 | 16 | 15
Not Completed | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: breast cancer survivors with known lymphedema
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.3) | 67.5 (10.3) | 66.0 (10.2) | 66.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 15 | 46
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 15 | 45
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 14 | 15 | 15 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 15 | 46
Time from surgery to lymphedema diagnosis [Median (Inter-Quartile Range); unit: months] | 7.2 [4 to 27] | 14.8 [5 to 108] | 30.0 [2 to 84] | 11.1 [3 to 73]
Duration of lymphedema prior to study enrollment [Median (Inter-Quartile Range); unit: months] | 27.0 [6 to 58] | 18.9 [5 to 73] | 25.2 [6 to 142] | 25.4 [6 to 86]

OUTCOME MEASURES:

1. Primary Outcome: LDex Change-
Description: Bioimpedance measured by units of LDex. As extracellular fluid accumulates (i.e. lymphedema develops) the LDex value increases.
Time Frame: Bioimpedance at baseline and end of treatment with the average number of treaments being 9 conducted over a median of up to 4 weeks.
Population: LDex units.
Measure: Median (Inter-Quartile Range); unit: LDex
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Number analyzed (Participants) | 15 | 16 | 15
LDex | 28.0 [17 to 35] | 17.8 [3 to 38] | 22.2 [11 to 37]

2. Secondary Outcome: Symptoms
Description: Yes/no response to a symptom listed on the Lymphedema Symptom Intensity and Distress Scale-Arm (LSIDS-A) self-report form.
Time Frame: Self report on last day of treatment with average treatments being 9 conducted over a median of up to 4 weeks.
Population: Total number of reported symptoms. Range of symptoms reported could be 0 to 36. Greater number of symptoms represents worse outcome.
Measure: Median (Inter-Quartile Range); unit: symptoms
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Number analyzed (Participants) | 15 | 16 | 15
symptoms | 12 [4 to 16] | 12.5 [6 to 16] | 14 [10 to 19]

3. Secondary Outcome: Quality of Life
Description: The Functional Assessment of Chronic Illness Therapy that measure quality of life -total score. Range of scores could be 0 to 148. Higher score represents higher quality of life.
Time Frame: Self-report on last day of treatment with average number of treatments being 9 conducted over a median of up to 4 weeks.
Measure: Median (Inter-Quartile Range); unit: total score
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Number analyzed (Participants) | 15 | 16 | 15
total score | 113.5 [100 to 129] | 116.25 [98 to 123] | 110 [102 to 123]

4. Primary Outcome: Whole Arm Volume Difference
Description: Whole arm measurement to determine volume.
Time Frame: Baseline and on last day of treatment with average number of treatments being 9 conducted over a median of up to 4 weeks.
Measure: Median (Inter-Quartile Range); unit: Whole Arm Volume % Difference
Groups:
- Mld Alone: therapist administered manual lymphatic drainage (mld)
  manual lymphatic drainage: therapist administered massage therapy
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Number analyzed (Participants) | 15 | 16 | 15
Whole Arm Volume % Difference | 15.0 [3 to 23] | 6.8 [0 to 17] | 13.4 [2 to 24]

ADVERSE EVENTS:
Time Frame: Participants were followed through the last treatment and there was an average of 9 treatments per group.
Groups:
- Laser Therapy Alone: therapist administered laser treatment
  laser: therapist administered laser
  No adverse events during the study.
- Mld Alone: therapist administered manual lymphatic drainage
  manual lymphatic drainage: therapist administered massage therapy
  No adverse events during the study.
- Laser and Mld Combined: therapist administered laser and mld
  Low Level Laser Therapy with Manual Lymphatic Drainage: therapist will give both mld and laser treatment
  No adverse events during the study.
Arm/Group | Laser Therapy Alone | Mld Alone | Laser and Mld Combined
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No